CLINICAL TRIAL: NCT05313659
Title: Intramuscular Ketamine Effect on Postnasal Surgery Agitation: a Double Blinded Randomized Controlled Trial.
Brief Title: Intramuscular Ketamine Effect on Postnasal Surgery Agitation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jordanian Royal Medical Services (Other)
Responsible Party: Principal Investigator, Husam A. Almajali, anesthesia specialist, Jordanian Royal Medical Services
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: postoperative agitation
Record Dates: First submitted 2022-03-20; First posted 2022-04-06 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Agitation, Emergence
Keywords: Agitation; Emergence; Ketamine; Intramuscular; Nasal surgery
MeSH Terms: conditions — Emergence Delirium; Psychomotor Agitation | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group-K (Experimental): At the end of surgery and immediately after the inhalational agent was discontinued, 2mL of normal saline containing 0.7 mg/kg racemic ketamine was administered intramuscularly to Group-K
  Interventions: Drug: Ketamine Hydrochloride
- group-S (No Intervention): At the end of surgery and immediately after the inhalational agent was discontinued, 2 mL of normal saline was administered intramuscularly.

INTERVENTIONS:
Drug: Ketamine Hydrochloride — intramuscular ketamine hydrochloride at dose of 0.7 mg/kg at the time of turning the inhalational agent off
  Arms: group-K

SUMMARY:
Emergence agitation (EA) is a common complication after nasal surgery. In this study, we aimed to investigate the effect of intramuscular ketamine on EA following septoplasty and open septorhinoplasty (OSRP) when administered at subanesthetic doses at the end of surgery. Sedation and Agitation scores were recorded using The Richmond agitation-sedation score after extubation.

DETAILED DESCRIPTION:
At the end of surgery and immediately after the inhalational agent was discontinued, 2mL of normal saline containing 0.7 mg/kg racemic ketamine was administered intramuscularly to Group-K, whereas 2 mL of normal saline was administered intramuscularly to Group-S using a 3 ml syringe. The injection site of both groups was at the lateral thigh. For postoperative analgesia, 0.07 mg/kg morphine was also given when turning off the inhalational agent. A nasal pack was used in all of the patients. The patients were ventilated with 100% oxygen at a flow rate of 7 L/min. Once the patients met the extubation criteria, they were extubated.

The EA level of the patients was evaluated immediately after extubation till the patient was handed over to the PACU using Richmond Agitation-Sedation Scale (RASS), Table 1, and the highest score was documented by the main investigators. In this study patients with a RASS score of +2 or more were considered to have EA.

ELIGIBILITY:
Inclusion Criteria:

1. Age group 18-64 years old
2. ASA I-II
3. BMI 20-29.9
4. Patients accepting the study and consenting
5. Undergoing general anesthesia for scheduled septoplasty or open septorhinoplasty.

Exclusion Criteria:

1. ketamine allergy
2. Morphine allergy
3. History of cardiac, neurological, or psychiatric disease, glaucoma,
4. Patients with a body mass index of less than 20 or more than 30 kg/m2

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 193 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-10-20 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Development of Agitation | immediately After extubation.
  Using The Richmond agitation-sedation score. The score being from(-5) to (+4) ; 2 and more being agitated patients and less than 2 not agitated.

CONTACTS AND LOCATIONS:
Overall Officials: Husam A. Almajali, MD, Principal Investigator — Jordanian Royal Medical Services; Ali M. Abu Dalo, MD, Principal Investigator — Jordanian Royal Medical Services
Locations (1):
- Jordanian Royal Medical Services, Amman, Jordan